CLINICAL TRIAL: NCT01373866
Title: Multimodal MRI-guided Repetitive Transcranial Magnetic Stimulation to Treat Drug-resistant Hallucinations: a Randomized Control Trial
Brief Title: Multimodal MRI-guided rTMS to Treat Refractory Hallucinations
Acronym: MULTIMODHAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009_17/0927; 2009-A00842-55 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2011-05-13; First posted 2011-06-15 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hallucinations; Schizophrenia; Perceptual Disorders
Keywords: Repetitive Transcranial Magnetic Stimulation; Neuronavigation; Functional Magnetic Resonance Imaging; Diffusion Tensor Imaging
MeSH Terms: conditions — Hallucinations; Schizophrenia; Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal MRI-guided rTMS (Experimental)
  Interventions: Device: MagPro X100 repetitive Transcranial Magnetic Stimulation
- Conventional T3-P3 rTMS (Active Comparator)
  Interventions: Device: MagPro X100 repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: MagPro X100 repetitive Transcranial Magnetic Stimulation — Target defined using both fMRI during hallucinations occurence and tractography.
  Parameters: 1 Hz/ 100% of the Motor Threshold/ 10 sessions (2/ day over 5 days)/ 1200 pulses/ session
  Arms: Multimodal MRI-guided rTMS
Device: MagPro X100 repetitive Transcranial Magnetic Stimulation — Target: T3-P3 (10-20 EEG international System). Parameters: 1 Hz/ 100% of the Motor Threshold/ 10 sessions (2/ day over 5 days)/ 1200 pulses/ session
  Arms: Conventional T3-P3 rTMS

SUMMARY:
* The efficacy of neuro-navigated rTMS for patients with schizophrenia suffering from drug-resistant multisensory hallucinations will be tested by the implementation of a double-blind randomized controlled trial (RCT)
* This study will use a combination of different MRI modalities (fMRI and DTI) to define with precision rTMS brain-targets in the case of multisensory hallucinations
* The investigators anticipate that multimodal MRI-guided rTMS will allow a significant improvement in the efficacy of neuromodulation treatment of refractory hallucinations

ELIGIBILITY:
Inclusion Criteria:

* Right-handed Female/Male, [13-60 y.o.],
* Schizophrenia (DSM-IV-TR diagnosis),
* Drug-resistant hallucinations (Kinon & Kane criteria, 1993),
* Unmodified antipsychotic dosage during the 30 days preceding rMTS,
* No anticonvulsive medication,
* No neurological disorder, no addictive behavior,
* Matched for sex, age and PANSS scores,
* Consent to participate to the study,

Exclusion Criteria:

* Pregnancy
* Contraindication to MRI scan
* Contraindication to rTMS treatment
* Claustrophobia
* No social insurance

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Severity and Frequency of Hallucinations | Assessed at baseline (t0) and longitudinally after the 10 rTMS sessions during the following month (D+15, M+1, M+3, M+6, M+12)
  Visual Analogue Scale (Severity)/ Visual Analogue Scale (Frequency rate)

SECONDARY OUTCOMES:
Clinical State | Assessed at baseline (t0) and longitudinally after the 10 rTMS sessions during the following month (D+15, M+1, M+3, M+6, M+12)
  Clinical Global Improvement [CGI]/ Positive & Negative Symptoms Scale [PANSS]/ Global Assessment of Functioning [GAF].
  For the auditory modality: Add the Auditory Hallucinations rating Scale [AHRS] frequency scale and total score/ Add the computerized Binary Scale of Auditory Speech Hallucinations [cbSASH]
MRI changes | Assessed at baseline (t0) and 1 month after the rTMS sessions (M+1)
  structural MRI/ functional MRI/ Diffusion Tensor Imaging/ MR-spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Jardri, M.D., Ph.D., Principal Investigator — Lille University Medical Centre, France
Locations (2):
- France (2):
  - Lille University Hospital Centre, Lille
  - Saint-Anne Psychiatric Hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demeulemeester M, Kochman F, Fligans B, Tabet AJ, Thomas P, Jardri R. Assessing early-onset hallucinations in the touch-screen generation. Br J Psychiatry. 2015 Mar;206(3):181-3. doi: 10.1192/bjp.bp.114.154153. PMID 25733569
- [Derived] Leroy A, Foucher JR, Pins D, Delmaire C, Thomas P, Roser MM, Lefebvre S, Amad A, Fovet T, Jaafari N, Jardri R. fMRI capture of auditory hallucinations: Validation of the two-steps method. Hum Brain Mapp. 2017 Oct;38(10):4966-4979. doi: 10.1002/hbm.23707. Epub 2017 Jun 28. PMID 28660668